CLINICAL TRIAL: NCT01701609
Title: Efficacy of a Cognitive Remediation Treatment in Adolescents With Schizophrenia Spectrum Disorders
Brief Title: Cognitive Remediation Therapy (CRT) in Adolescents With EOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Centro de Investigación Biomédica en Red de Salud Mental (Network)
Responsible Party: Principal Investigator, Olga Puig, Olga Puig Navarro, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI07/90054; ETES07/90054 (Other Grant/Funding Number: ISCIII)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
Keywords: early-onset schizophrenia; adolescents; cognition; cognitive remediation therapy
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Remediation Therapy (Experimental): CRT: Frontal/Executive Program. The program has a duration of 40 sessions, with two session for week. Is is carried out individually and utilizes paper and pencil tasks. The main technique utilized is the scaffolding in a context of learning without errors.
  Interventions: Behavioral: Cognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy
  Other Names: Cognitive training; Cognitive enhancement

SUMMARY:
Cognitive Remediation Therapy (CRT) can enhance cognitive performance in schizophrenia improving functional outcome. But most of the studies have involved participants who are in average in their mid 30s, and little is known about the efficacy of CRT in adolescents with early-onset schizophrenia (EOS). The aim of this study is to investigate efficacy of CRT in improving cognitive performance and functional outcome in adolescents with EOS. We expect to find that CRT improves cognitive and functional outcomes in adolescents with schizophrenia.

DETAILED DESCRIPTION:
Early-onset schizophrenia (EOS) is associated with worse course and poor outcome than adulthood schizophrenia. Cognitive deficits are known to be a core feature in EOS, with large deficits on almost all cognitive domains. Importantly, cognitive deficits are known to be strong predictors of psychosocial and functional outcomes in schizophrenia and also in the early-onset form of the illness. Cognitive Remediation Therapy (CRT) is a behavioral training based intervention that aims to improve cognitive processes (attention, memory, executive function, social cognition or metacognition) with the goal of durability and generalization. It has been demonstrated that CRT improve cognitive deficits and functional outcome in adult patients but there are very few studies with adolescent samples.

A controlled randomized study will be carry out with two groups: patients receiving treatment as usual plus CRT, and patients receiving treatment as usual (TAU). The independent variable is the cognitive remediation treatment. The CRT will be applied according to the manual of Wykes and Reeder (2005). The program has a duration of 40 sessions, with two session for week. It is carried out individually and utilizes paper and pencil tasks. The main technique utilized is the scaffolding in a context of learning without errors.

The main dependent variable is the cognitive performance measured through neuropsychological tests. Other secondary dependent variables are functional outcome and clinical symptoms obtained from the psychometric evaluation.

All participants will be evaluated before and after the experimental intervention in several neurocognitive domains, clinical symptoms and functional outcome. The evaluations will be carried out by expert evaluators. Intention-to-treat analysis will be carry out using the statistical package SPSS v 18.

ELIGIBILITY:
Inclusion Criteria:

* age between 12 and 18 years
* a DSM-IV-TR schizophrenia-type disorder (schizophrenia or schizoaffective disorder), with onset before the age of 17
* being clinically and pharmacologically stabilized during the last 6 weeks before the baseline assessment
* the estimation of not modifying pharmacological antipsychotic treatment
* presence of cognitive deficit confirmed by the neuropsychological battery

Exclusion Criteria:

* IQ below 70
* presence of an active misuse disorder
* presence of organic brain syndromes or neurological disorders
* having received electroconvulsive therapy in the previous 6 months

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 20 weeks
  Change from baseline in neuropsychological test scores of memory, executive functions, working memory and processing speed at post-treatment evaluation

SECONDARY OUTCOMES:
Functional outcome | 20 weeks
  Change in real-world functioning scales, self-esteem and caregiver burden at post-treatment evaluation
Symptoms | 20 weeks
  Change from baseline in measures of clinical symptoms at post-treatment evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Olga Puig, PhD, Principal Investigator — Hospital Clinic of Barcelona; Rafael Penadés, PhD, Study Director — Hospital Clinic of Barcelona; Josefina Castro-Fornieles, MD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Department of Child and Adolescent Pyshicatry and Psychology, Barcelona, Catalonia, Spain

REFERENCES:
- [Result] Puig O, Penades R, Baeza I, De la Serna E, Sanchez-Gistau V, Bernardo M, Castro-Fornieles J. Cognitive remediation therapy in adolescents with early-onset schizophrenia: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Aug;53(8):859-68. doi: 10.1016/j.jaac.2014.05.012. Epub 2014 Jun 21. PMID 25062593